CLINICAL TRIAL: NCT03052257
Title: Improving Glaucoma Medication Adherence
Brief Title: Improve Glaucoma Medication Adherence
Acronym: MAGIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 15-113
Record Dates: First submitted 2017-01-18; First posted 2017-02-14 (Actual); Results first posted 2020-08-27 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Glaucoma
Keywords: Glaucoma; Disease management; Smart bottle
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants will be randomized to receive either a general eye health educational session (control arm) or an educational intervention developed to improve glaucoma medication adherence (intervention arm). All participants will be provided with a "smart bottle" to house one of their glaucoma medications. The smart bottle records the date and time that the bottle is opened.
  Interventions: Behavioral: Educational - glaucoma; Behavioral: Dose monitoring and reminder
- Control (Active Comparator): Participants will be randomized to receive either a general eye health educational session (control arm) or an educational intervention developed to improve glaucoma medication adherence (intervention arm). All participants will be provided with a "smart bottle" to house one of their glaucoma medications. The smart bottle records the date and time that the bottle is opened.
  Interventions: Behavioral: Educational - general; Behavioral: Dose monitoring

INTERVENTIONS:
Behavioral: Educational - glaucoma — Discussion of glaucoma and the potential for blindness, facilitated by the glaucoma educator using a 3-dimensional model eye and photographic representation of glaucomatous vision loss; One-one-one demonstration of eye drop instillation techniques, Provision of a mnemonic aid which alerts the participant to missed doses; Review of the participant manual: An illustrated brochure on glaucoma and eye drop instillation. An individualized schedule for dosing of glaucoma medications. Individualized suggestions for improving adherence based on the subject's responses to the (SASES).
  Arms: Intervention
Behavioral: Dose monitoring and reminder — Participants will be provided with a "smart bottle" to house one of their glaucoma medications. The smart bottle records the date and time that the bottle is opened. For participants in the intervention arm only, a reminder through AdhereTech will be activated.
  Other Names: Smart bottle reminder
  Arms: Intervention
Behavioral: Educational - general — The control information session will include review of a Powerpoint presentation on general eye health, including but not specific to glaucoma.
  Arms: Control
Behavioral: Dose monitoring — Participants will be provided with a "smart bottle" to house one of their glaucoma medications. The smart bottle records the date and time that the bottle is opened.
  Other Names: Smart bottle
  Arms: Control

SUMMARY:
The proposed study is a randomized controlled trial enrolling Veterans with medically treated glaucoma who report less than 100% adherence to the prescribed glaucoma therapy. Participants will be randomized to receive either a one-on-one session with a member of the research team discussing the disease process and strategies for administering eye drops (intervention) or a one-on-one session with a member of the research team discussing general eye health (control). All participants will be provided with a "smart bottle" to house their glaucoma medications. The smart bottle records the date and time that the bottle is opened. For participants in the intervention arm only, a reminder function will be activated. The proportion or prescribed doses taken according to the monitor will be compared for the two groups.

DETAILED DESCRIPTION:
The purpose if this study is to improve glaucoma medication adherence in Veterans with medically-treated glaucoma. The study design is a single-site randomized controlled trial. Specific Aim 1. Evaluate the impact of an intervention to improve glaucoma medication adherence among Veterans at 6-month follow up.

Hypothesis 1: Veterans randomized to the intervention will have a greater proportion of prescribed glaucoma medication doses taken as measured by the electronic medication monitor in the 6 months following the intervention compared to Veterans randomized to the control arm.

The primary outcome for hypothesis 1A is the proportion of prescribed doses taken according to the electronic monitor. Participants in both arms will receive the electronic monitor or "smart bottle," which wirelessly transmits the date and time of opening of the smart bottle to the study team. From these medication events, the proportion of prescribed doses will be derived, defined as the ratio of the number of times the smart bottle was opened to the required number of doses prescribed according to the medical record over the period of time that the bottle is in use. For example, if a participant is advised to take his or her glaucoma drop twice a day for the 180 days that the bottle is in use and the smart bottle reveals 135 openings over the same time period, the proportion of prescribed doses taken is 37.5%.

Specific Aim 2. Evaluate the impact of the intervention on intensification of glaucoma therapy among Veterans at 12-month follow-up.

Hypothesis 2: The proportion of Veterans in the intervention arm that are prescribed more intensive glaucoma therapy, defined as addition of adjuvant glaucoma medication or recommendation for laser or glaucoma surgery will be less than the proportion of Veterans in the control arm who are prescribed more intensive glaucoma therapy in the 12 months following the intervention.

Baseline data collection will include cataloging the current glaucoma medication regimen prescribed to the participant. Chart abstractions will be performed at 12 months following the baseline visit and intensification of glaucoma therapy will be defined as either 1) the addition of another glaucoma medication to the baseline regimen, 2) recommendation for glaucoma laser treatment, or 3) recommendation for glaucoma surgery in the 12 months following the baseline visit . The investigators will collect these data at 12 months because the Metrics study suggested that 55% of participants in the control arm will have intensification of therapy within one year.

Specific Aim 3. Evaluate the incremental cost-effectiveness and budget and workflow impacts of the intervention compared to usual care.

Hypothesis 3: The intervention will be cost-effectiveness for the following ratios: 1) cost per percentage improvement in medication adherence; 2) cost per blindness averted; and 3) cost per quality-adjusted-life years saved.

A direct measurement approach will be used to estimate per-patient intervention and control arm costs. Glaucoma-related health care utilization costs will be derived from VA administrative datasets. The cost estimates will be combined with observed improvement in medication adherence and reduction in escalation in therapy to estimate the first two incremental cost effectiveness ratios. Simulation using Markov modeling will be used to estimate the incremental cost per blindness averted and quality-adjusted life years (QALYs) gained. Cost estimates and labor time data collected will be combined with glaucoma prevalence rates among Veterans to estimate overall budget and workload impacts to the VA healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma [primary open angle glaucoma, pigment dispersion glaucoma, pseudoexfoliation glaucoma, combined mechanism glaucoma, low tension glaucoma] recorded in the medical record
* Prescribed glaucoma eye drops,
* Visual field performed within the last 9 months.

  * As visual field testing is standard care glaucoma and the investigators wish to establish baseline glaucoma severity, the investigators will require that subjects have a visual field test documented in the chart within 9 months of enrollment.

Exclusion Criteria:

Exclusion criteria for patients At Screener:

* "How confident are you that you always remember to use your glaucoma medications?"

  * not at all confident
  * somewhat confident
  * very confident)
* And "In the past 4 weeks, did you ever forget to take your medicine?"

  * Veterans who respond both "very confident" and "no", respectively, will be excluded

Inclusion criteria for companions at screener:

* Willing to participate in assisting the patient with glaucoma drops and
* Willing to accompany the patient to the intervention visit for participants in the intervention arm or eye health education visit for participants in the control arm.

Exclusion criteria for companions: Unable or unwilling to attend baseline visit and intervention or control arm educational session with patient participant.

Exclusion criteria for patients or companions:

* Lacks proficiency in English,
* Lacks either a cell phone or landline phone.

Exclusion criteria for patients post randomization:

* Decision by patient and provider to cease glaucoma medication use
* Change in functional status such that the drops are no longer administered by the patient or the companion (such as nursing home care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly W. Muir, MD MHSc, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Hein AM, Rosdahl JA, Bosworth HB, Woolson SL, Olsen MK, Kirshner MA, Muir KW. The Association of an Upper Extremity Functional Survey and Glaucoma Medication Administration Success. Curr Eye Res. 2019 Oct;44(10):1150-1156. doi: 10.1080/02713683.2019.1625405. Epub 2019 Jun 11. PMID 31157555
- [Result] Rosdahl JA, Hein AM, Bosworth HB, Woolson S, Olsen M, Kirshner M, Hung A, Muir KW. Randomized controlled trial of an education-based intervention to improve medication adherence: Design considerations in the medication adherence in glaucoma to improve care study. Clin Trials. 2021 Jun;18(3):343-350. doi: 10.1177/1740774520988291. Epub 2021 Jan 25. PMID 33487050
- [Result] Muir KW, Rosdahl JA, Hein AM, Woolson S, Olsen MK, Kirshner M, Sexton M, Bosworth HB. Improved Glaucoma Medication Adherence in a Randomized Controlled Trial. Ophthalmol Glaucoma. 2022 Jan-Feb;5(1):40-46. doi: 10.1016/j.ogla.2021.04.006. Epub 2021 Apr 20. PMID 33892170
- [Result] Williams AM, Theophanous C, Muir KW, Rosdahl JA, Woolson S, Olsen M, Bosworth HB, Hung A. Within-Trial Cost-Effectiveness of an Adherence-Enhancing Educational Intervention for Glaucoma. Am J Ophthalmol. 2022 Dec;244:216-227. doi: 10.1016/j.ajo.2022.08.011. Epub 2022 Aug 21. PMID 36002073
- [Result] Buehne KL, Rosdahl JA, Hein AM, Woolson S, Olsen M, Kirshner M, Sexton M, Bosworth HB, Muir KW. How Medication Adherence Affects Disease Management in Veterans with Glaucoma: Lessons Learned from a Clinical Trial. Ophthalmic Res. 2023;66(1):489-495. doi: 10.1159/000528857. Epub 2023 Jan 5. PMID 36603568
- See also: Intervention Arm Content Video testimonial from a glaucoma patient — http://www.eyecareamerica.org/news/press/

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Participants were randomized educational intervention developed to improve glaucoma medication adherence. This included a discussion of glaucoma and the potential for blindness, facilitated by the glaucoma educator using a 3-dimensional model eye and photographic representation of glaucomatous vision loss; One-one-one demonstration of eye drop instillation techniques, provision of a mnemonic aid which alerts the participant to missed doses; Review of the participant manual: An illustrated brochure on glaucoma and eye drop instillation, an individualized schedule for dosing of glaucoma medications. Individualized suggestions for improving adherence based on the subject's responses to the (SASES). Participants were provided with a "smart bottle" to house one of their glaucoma medications. The smart bottle recorded the date and time that the bottle was opened and a reminder through AdhereTech was activated.
- Control: Participants randomized to receive general eye health educational session, the control information session included review of a PowerPoint presentation on general eye health, including but not specific to glaucoma. All participants were provided with a "smart bottle" to house one of their glaucoma medications. The smart bottle recorded the date and time that the bottle is opened.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 100 | 100
Completed | 95 | 97
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (8.6) | 67.1 (8.1) | 67.5 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 96 | 91 | 187
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 14
  Not Hispanic or Latino | 90 | 96 | 186
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 66 | 73 | 139
  White | 30 | 21 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 100 | 200
Doses Per Day of Monitored Medication [Count of Participants; unit: Participants] — Participants will be randomized at the first informational session in a 1:1 allocation to the intervention or to the control arm. Randomization will be stratified according to if a companion is or is not enrolled in the study with the participant and according to whether the glaucoma medication housed by the AdhereTech bottle is prescribed to be take once daily or more than once daily.
  Participants
    One Dose Per Day | 44 | 43 | 87
    More Than One Dose Per Day | 56 | 57 | 113
Companion Status [Count of Participants; unit: Participants] — Participants will be randomized at the first informational session in a 1:1 allocation to the intervention or to the control arm. Randomization will be stratified according to if a companion is or is not enrolled in the study with the participant and according to whether the glaucoma medication housed by the AdhereTech bottle is prescribed to be take once daily or more than once daily.
  Participants
    Companion at Randomization | 20 | 21 | 41
    No Companion at Randomization | 80 | 79 | 159

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Prescribed Glaucoma Medication Doses Taken on Schedule
Description: Will veterans randomized to the intervention have a greater proportion of prescribed glaucoma medication doses taken as measured by the electronic medication monitor in the 6 months following the intervention compared to Veterans randomized to the control arm? The electronic bottle records the date and time that the bottle is opened. For participants in the intervention arm only, a reminder through the electronic bottle will be activated. The outcome measure is the proportion of prescribed doses taken with a minimum of Zero and a maximum of One; where higher scores indicate more adherence.
Time Frame: Randomization to 6 Months
Population: 95 Intervention: Of the 100 randomized to Intervention - 2 subjects withdrew after randomization and 3 subjects excluded for not having at least 25 weeks of adherence data 97 Control: Of the 100 randomized to Control - 1 subject excluded by PI for not taking medication and 2 subjects excluded for not having at least 25 weeks of adherence data
Measure: Least Squares Mean (95% Confidence Interval); unit: proportion of doses
Arm/Group | Intervention | Control
Number analyzed (Participants) | 95 | 97
proportion of doses | .84 [0.78 to 0.90] | 0.62 [0.56 to 0.67]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.0001, Regression, Linear; Median Difference (Final Values) = 0.23, 95% CI 2-sided [0.15 to 0.30], Standard Error of Mean 0.04

2. Secondary Outcome: VA Medical Resource Use and Costs
Description: The investigators will investigate the overall budget impacts to the VA healthcare system. The main intervention costs are labor inputs, consisting of the one-time fixed labor cost of training and the variable labor cost of conducting the adherence intervention. The VA healthcare system also incurs costs, such as administration, utilities, and custodial services that cannot be directly attributed to a given health care service but nonetheless should be included in the cost analysis.
Time Frame: 6 months
Population: 100 Intervention 100 Control
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | Intervention | Control
Number analyzed (Participants) | 100 | 100
USD | 10947 (19341) | 12939 (25199)

3. Other Pre Specified Outcome: Number of Participants With Newly Prescribed Glaucoma Therapy
Description: Will the proportion of Veterans in the intervention arm that are prescribed more intensive glaucoma therapy be less than the proportion of Veterans in the control arm who are prescribed more intensive glaucoma therapy in the 12 months following the intervention? Baseline data collection will include cataloging the current glaucoma medication regimen prescribed to the participant. Chart abstractions will be performed at 12 months following the baseline visit and intensification of glaucoma therapy will be defined as either 1) the addition of another glaucoma medication to the baseline regimen, 2) recommendation for glaucoma laser treatment, or 3) recommendation for glaucoma surgery in the 12 months following the baseline visit .
Time Frame: 12 Months
Population: 200 randomized Veterans who are patients of the Durham VA Eye Clinic with medically-treated glaucoma.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 100 | 100
Participants | 23 | 24

4. Other Pre Specified Outcome: Total Cost at 6 Months
Description: The proportion of participants attaining equal or >80% adherence as measured by electronic monitor, total intervention and medical resource costs, and incremental cost effectiveness ratios comparing intervention to control at 6 months.
Time Frame: 6 months
Population: 100 Intervention (hypothetical cohort) 100 Control (hypothetical cohort)
Measure: Number; unit: USD
Arm/Group | Intervention | Control
Number analyzed (Participants) | 100 | 100
USD | 1,149,600 | 1,298,700

5. Other Pre Specified Outcome: VA Healthcare Workflow Effectiveness
Description: The investigators will investigate the overall workload impacts to the VA healthcare system. Cost estimates and labor time data collected will be combined with glaucoma prevalence rates among Veterans to estimate overall workload impacts to the VA healthcare system.
Time Frame: 12 months
Population: Workflow changed significantly over the course of the study such that this outcome became not feasible to assess. Over the time that participants were enrolled, we had multiple staff and doctor changes, not to mention the pandemic.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Cost-effectiveness Compared to Usual Care for Cost Per Blindness Averted
Description: Will the intervention be cost-effectiveness compared to usual care for cost per blindness averted
Time Frame: 12 months
Population: While the long-term goal of this research program is to reduce glaucoma-related blindness in Veterans; in the course of the study period no participants went blind. We were unable to calculate this hypothesized outcome.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Within-Trial Cost-Effectiveness of Adherence
Description: Will the intervention be cost-effectiveness compared to usual care? Total cost was calculated by adding the mean medical resource cost per patient to the cost of the intervention ($549) or the control ($48), then multiplying the total by the number of patients per group (100)
Time Frame: 6 months
Measure: Number; unit: USD
Arm/Group | Intervention | Control
Number analyzed (Participants) | 100 | 100
USD | 1,149,600 | 1,298,700

8. Other Pre Specified Outcome: VA Workflow Effectiveness
Description: The investigators will investigate the overall workload impacts to the VA healthcare system.
Time Frame: 12 months
Population: as for outcome 5
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 4/100 | 2/100
Serious Adverse Events (participants affected / at risk) | 3/100 | 2/100
Other Adverse Events (participants affected / at risk) | 1/100 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=100) | Control (N=100)
Death (General disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=100) | Control (N=100)
Hospitalization (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT03052257/Prot_SAP_000.pdf